CLINICAL TRIAL: NCT02853877
Title: Translating Insights From Behavioral Economics and Self-Determination Theory to Promote Sustained Weight Loss Among Obese Employees
Brief Title: Helping Employees Lose Pounds
Acronym: HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey T. Kullgren, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00107647
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Incentive (Experimental): Participants in the Weekly Incentive arm will be asked to weigh in each week during a 12 week intervention period. They will receive tailored messages and have an opportunity to win a financial reward each week they meet their weight loss goal. Participants will be asked to complete a final weight measurement at week 24.
  Interventions: Behavioral: Weekly Incentive
- Weekly Weigh-In (No Intervention): Participants in the Weekly Weigh-In arm will be asked to weigh in each week during a 12 week intervention period. Participants will be asked to complete a final weight measurement at week 24.

INTERVENTIONS:
Behavioral: Weekly Incentive — The tailored incentives intervention aims to assess the impact of tailored messaging and financial incentives on weight loss among obese employees.
  Arms: Weekly Incentive

SUMMARY:
This study will evaluate the effectiveness of financial incentives and messaging tailored to individual goals and aspirations to promote and sustain weight loss. This is a 2-arm randomized controlled trial that will recruit eligible employees at a large university to participate in a 3-month weight loss program, followed by a 3-month follow-up period. The primary outcome will be change in autonomous motivation for weight loss.

The study hypothesis is that intervention group participants will have a greater increase in autonomous motivation for weight loss than participants in the control group at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Interested in losing weight
* Body Mass Index between 30 and 40 kg/m2
* Have wireless internet at home
* Have Android or iOS smart device
* Willing to record themselves weighing in on a scale or let a family member record them weighing in on a scale

Exclusion Criteria:

* Pregnant or lactating, or intending to become pregnant in the next 6 months
* Taking medication (other than metformin) for diabetes to control blood sugar
* Having a serious psychiatric diagnosis, unstable medical conditions or experienced a heart attack or stroke in the past 6 months
* Having a history of drug or alcohol abuse or addiction to prescription medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Change in autonomous motivation as measured by the Treatment Self-Regulation Questionnaire | 12 weeks

SECONDARY OUTCOMES:
Change in weight as measured by participant weight measurements using Withings scales | 12 weeks and 24 weeks

OTHER OUTCOMES:
Change in autonomous motivation as measured by the Treatment Self-Regulation Questionnaire | 24 weeks
Change in physical activity as measured by the short form of the International Physical Activity Questionnaire | 12 weeks and 24 weeks
Change in eating behaviors as measured by the Three Factor Eating Questionnaire | 12 weeks and 24 weeks
Change in participation in weight-related wellness programs as measured by responses to the question "In the past 3 months, have you participated in any health and wellness programs?" | 12 weeks and 24 weeks
Change in self-efficacy to lose weight as measured by the Perceived Competence Scale | 12 weeks and 24 weeks
Change in stage of change for weight loss as measured by responses to the questions "Are you currently trying to lose weight?" and "Do you intend to try to lose weight in the near future?" | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T Kullgren, MD,MS,MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No